CLINICAL TRIAL: NCT01512446
Title: Comparison of the Effect of an Ongoing Treatment With Alendronate or a Drug Holiday on the Fracture Risk in Osteoporotic Patients With Bisphosphonate Long Term Therapy
Acronym: BILANZ
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Evangelisches Krankenhaus Lutherhaus gGmbH (Industry)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. med. Johannes Pfeilschifter, Head of Department of Internal Medicine III, Evangelisches Krankenhaus Lutherhaus gGmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011.1.42; 2011-000290-31 (EudraCT Number)
Record Dates: First submitted 2012-01-11; First posted 2012-01-19 (Estimated); Results first posted 2019-01-17 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Osteoporotic fractures; Bisphosphonate; Pretreatment with bisphosphonates
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alendronate (Active Comparator)
  Interventions: Drug: Alendronate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alendronate — 70 mg per week
  Other Names: Fosamax
  Arms: Alendronate
Drug: Placebo — 1 pill per week
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of bisphosphonates in long term treatment of osteoporosis.

DETAILED DESCRIPTION:
Is a continued treatment with alendronate for another two years after a preceding therapy with bisphosphonates of at least four years able to reduce the incidence of new osteoporotic fractures in patients at high fracture risk compared to a therapy-free interval?

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women or men > 60 years
* DXA T-Score at lumbar spine, total hip or femur neck <-2,0 before the start of the bisphosphonate therapy or at baseline or at least one low trauma vertebral fracture grade 2-3 or multiple low trauma vertebral fractures independent of bone mineral densitiy
* Pretreatment with bisphosphonates for at least four years
* Risk for hip and vertebral fractures min. 30% according to DVO-guideline for osteoporosis 2009
* Signed informed consent

Exclusion Criteria:

* Other pharmacological treatment of osteoporosis during the last 48 months
* Other bone diseases
* Malabsorption syndromes
* Renal insufficiency with a calculated creatinine clearance < 35 ml/min
* Diseases of the esophagus, delayed esophageal clearance
* UUnability to realise the intake instructions
* Hypocalcemia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Pfeilschifter, Prof. Dr. med., Study Director — Alfried Krupp Krankenhaus Essen Steele
Locations (1):
- Department of Internal Medicine III, Alfried Krupp Krankenhaus Essen Steele, Essen, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was early terminated due to a low recruitment rate
Groups:
- Placebo: Placebo, administered orally once weekly
- Alendronate: Alendronate 70 mg, administered orally once weekly
Period: Overall Study
Arm/Group | Placebo | Alendronate
Started | 221 | 215
Safety Analysis Set (Received at least one dose of study medication) | 197 | 188
Completed | 0 | 0
Not Completed | 221 | 215

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alendronate | Total
Number analyzed (Participants) | 221 | 215 | 436
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.3 (6.9) | 74.3 (7.1) | 74.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 203 | 397
  Male | 27 | 12 | 39
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 221 | 215 | 436

OUTCOME MEASURES:

1. Primary Outcome: Number of New Osteoporotic Fractures
Description: Number of new osteoporotic fractures. All fractures which occurred without high impact trauma (i.e. atraumatically, minor accidents and falls from standing height and lower) were regarded as osteoporotic fractures, except for fractures of fingers, face, skull and toes.
Time Frame: From baseline to study termination (mean duration 5.6 months)
Population: Full Analysis Set (all randomized participants)
Measure: Number; unit: osteoporotic fractures
Arm/Group | Placebo | Alendronate
Number analyzed (Participants) | 221 | 215
osteoporotic fractures | 5 | 5

2. Secondary Outcome: Mortality
Description: Number of deaths
Time Frame: From baseline to study termination (mean duration 5.6 months)
Population: Full Analysis Set (all randomized participants)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Alendronate
Number analyzed (Participants) | 221 | 215
Participants | 2 | 0

3. Secondary Outcome: Combination of New Osteoporotic Fractures and Deaths
Description: Number of participants with a new osteoporotic fracture or death
Time Frame: From baseline to study termination (mean duration 5.6 months)
Population: Full Analysis Set (all randomized participants)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Alendronate
Number analyzed (Participants) | 221 | 215
Participants | 7 | 5

ADVERSE EVENTS:
Arm/Group | Placebo | Alendronate
Serious Adverse Events (participants affected / at risk) | 38/197 | 31/188
Other Adverse Events (participants affected / at risk) | 113/197 | 94/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=197) | Alendronate (N=188)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreas infection (Gastrointestinal disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Atypical femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 — toe fracture
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 2 — knowledge about one fractured sacrum was obtained post-study.
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 1 — 1 pelvic fracture occurred within 30 days after study termination
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 2 — 1 high impact fracture
Catheterisation cardiac (Investigations) | 1 | 0
Hysteroscopy (Investigations) | 0 | 1
Anaemia vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Sciatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Angioplasty (Surgical and medical procedures) | 1 | 0
Aortic valve replacement (Surgical and medical procedures) | 1 | 0
Dupuytren's contracture operation (Surgical and medical procedures) | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 2 | 0
Peripheral artery angioplasty (Surgical and medical procedures) | 1 | 0
Salpingo-oophorectomy (Surgical and medical procedures) | 0 | 2
Shoulder operation (Surgical and medical procedures) | 0 | 1
Toe operation (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0
Haematoma infection (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 2
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=197) | Alendronate (N=188)
Abdominal pain upper (Gastrointestinal disorders) | 23 | 15
Constipation (Gastrointestinal disorders) | 23 | 11
Tooth disorder (Gastrointestinal disorders) | 11 | 9
Fatigue (General disorders) | 30 | 27
Hyperhidrosis (General disorders) | 30 | 21
Oedema peripheral (General disorders) | 19 | 14
Upper respiratory tract infection (Infections and infestations) | 21 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 | 44
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 39 | 27
Dizziness (Nervous system disorders) | 38 | 22
Headache (Nervous system disorders) | 22 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 14
Cutaneous symptom (Skin and subcutaneous tissue disorders) | 21 | 14
Hypertension (Vascular disorders) | 23 | 13

LIMITATIONS AND CAVEATS:
Due to a low recruitment rate, the study was early terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes